CLINICAL TRIAL: NCT02924844
Title: Impact of the Implementation of a Clinical Pharmacy Bundle on Intensive Care Unit Patient Outcomes and Cost Expenditures
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 14/05.03
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Intensive Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Observation period before presence of clinical pharmacist: The group of patients was observed between Janary 2013 and December 2013
- Period with presence of clinical pharmacist: The group of patients was observed between January 2014 and June 2015.

SUMMARY:
The aim of this before-after study was to assess the impact of a clinical pharmacy bundle of care activities on patient outcomes (length of hospital stay as a primary endpoint) and cost expenditure in two French ICUs.

ELIGIBILITY:
Inclusion Criteria:

* Intensive Care Unit patients on weekdays

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The two study populations are composed of all patients present in the ICU on weekdays.
  The first population is composed of patients present between January 2013 and December 2013.
  The second population is composed of patients present between January 2014 and June 2015.
Sampling Method: Probability Sample
Enrollment: 2787 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | expected average of 20 days

SECONDARY OUTCOMES:
Intensive Care Unit length of stay | Expected maximum of 10 days
Mechanical ventilation duration | Expected maximum of 10 days
Intensive care unit mortality rate | Expected maximum of 10 days
Hospital mortality rate | End of hospital stay (expected average of 20 days)
Patient cost expenditure | End of hospital stay (expected average of 20 days)

OTHER OUTCOMES:
The rate of isolation of multidrug resistant organisms | End of hospital stay (expected average of 20 days)